CLINICAL TRIAL: NCT06736912
Title: A Randomized, Double-blind, Placebo-controlled, Single/multiple Dosing, Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety/tolerability, Pharmacokinetic/pharmacodynamic Characteristics and Food Effect After Oral Administration of IN-114199 in Healthy Participants
Brief Title: This Study Aims to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties and Food Effect of IN-114199 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IN_IBA_102
Record Dates: First submitted 2024-11-25; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Chronic Idiopathic Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part I(Cohort I) IN-114199 2.5 mg or Placebo (Experimental): SAD
  Interventions: Drug: IN-114199 2.5mg or placebo
- Part I(Cohort 2) IN-114199 5 mg or Placebo (Experimental): SAD and FES
  Interventions: Drug: IN-114199 5mg or placebo
- Part I(Cohort 3) IN-114199 10 mg or Placebo (Experimental): SAD and FES
  Interventions: Drug: IN-114199 10mg or placebo
- Part I(Cohort 4) IN-114199 20 mg or Placebo (Experimental): SAD and FES
  Interventions: Drug: IN-114199 20mg or placebo
- Part I(Cohort 5) IN-114199 40 mg or Placebo (Experimental): SAD
  Interventions: Drug: IN-114199 40mg or placebo
- Part II(Cohort I) IN-114199 2.5 mg or Placebo (Experimental): MAD
  Interventions: Drug: IN-114199 2.5mg or placebo
- Part II(Cohort 2) IN-114199 5 mg or Placebo (Experimental): MAD
  Interventions: Drug: IN-114199 5mg or placebo
- Part II(Cohort 3) IN-114199 10 mg or Placebo (Experimental): MAD
  Interventions: Drug: IN-114199 10mg or placebo
- Part II(Cohort 4) IN-114199 20 mg or Placebo (Experimental): MAD
  Interventions: Drug: IN-114199 20mg or placebo

INTERVENTIONS:
Drug: IN-114199 2.5mg or placebo — IN-114199 2.5mg or placebo (1 Tablet, QD)
  Arms: Part I(Cohort I) IN-114199 2.5 mg or Placebo; Part II(Cohort I) IN-114199 2.5 mg or Placebo
Drug: IN-114199 10mg or placebo — IN-114199 10mg or placebo (1 Tablet, QD)
  Arms: Part I(Cohort 3) IN-114199 10 mg or Placebo; Part II(Cohort 3) IN-114199 10 mg or Placebo
Drug: IN-114199 20mg or placebo — IN-114199 10mg or placebo (2 Tablets, QD)
  Arms: Part I(Cohort 4) IN-114199 20 mg or Placebo; Part II(Cohort 4) IN-114199 20 mg or Placebo
Drug: IN-114199 40mg or placebo — IN-114199 10mg or placebo (4 Tablets, QD)
  Arms: Part I(Cohort 5) IN-114199 40 mg or Placebo
Drug: IN-114199 5mg or placebo — IN-114199 2.5mg or placebo (2 Tablets, QD)
  Arms: Part I(Cohort 2) IN-114199 5 mg or Placebo; Part II(Cohort 2) IN-114199 5 mg or Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic properties and food effect of IN-114199 in healthy participants

DETAILED DESCRIPTION:
Part A: SAD and FES study

* To evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic properties of a single oral dose of IN-114199 in healthy adults
* To compare and evaluate the effects of food on the safety, tolerability, pharmacokinetic and pharmacodynamic properties of a single oral dose of IN-114199 in healthy adults

Part B: MAD study

- To evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic properties of repeated oral doses of IN-114199 in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 years and ≤ 63 years on the date of the written informed consent
* Healthy subjects were defined as individuals who defecated almost every day for ≥ 6 months
* Body weight of ≥ 40.0 kg and ≤ 100.0 kg, with body mass index (BMI) of ≥ 18.5 kg/m2 and ≤ 29.9 kg/m2 at the time of screening
* Those who have fully understood this clinical trial via detailed explanation, were willing to voluntarily participate in this study, and agreed to give written informed consent prior to the screening procedure.
* Those who are judged eligible for this study upon judgment of the investigator in screening tests established depending on the characteristics of investigational product (examinations by interview, clinical laboratory test, physical examinations, etc.).

Exclusion Criteria:

* Presence or history of clinically significant liver, kidney, nervous system, respiratory system, endocrine system, blood and tumor, cardiovascular system, urinary system or psychiatric disease
* Presence or history of gastrointestinal disorder (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) that may influence the safety and pharmacodynamic assessments of the investigational product and history of gastrointestinal surgery (except simple appendectomy and hernia surgery), hemostatic disorder or hemorrhage-related disease
* Hypersensitivity to drugs including the ingredients of the investigational product and other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity
* Positive result in serology tests (Hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test)
* Subjects who have history of drug abuse, or who have a positive urine test for drugs of abuse.
* Blood AST(SGOT), and ALT(SGPT) > 60 IU/L at the screening test
* Showing the following findings on ECG at the screening test: QT > 480 msec(all), QTcB>450(male), QTcB>470(female)
* Subjects who have taken any drugs known to significantly induce (e.g., barbiturates) or inhibit drug-metabolizing enzymes within 1 month prior to the expected initial application date.
* Subjects who have participated in other clinical trials within 6 months prior to the expected initial application date
* Subjects who have history of regular alcohol consumption exceeding 21 units/week (1 unit = 10 g = 12.5 mL of pure alcohol) or subjects who cannot avoid drinking alcohol from 3 days prior to the expected initial application date to the discharge
* Subjects who have history of average use of 10 cigarettes daily
* Subjects who consumed caffeine-containing food (coffee, green tea, black tea, carbonated beverage, coffee-flavored milk, tonics, etc.) or subjects who cannot avoid drinking caffeine-containing food from 3 days prior to the expected initial application date to the discharge
* Subjects are unable to use a highly effective method of contraception (e.g., correctly placed intrauterine device(IUD), sterilization surgery (vasectomy, tubal ligation, etc.))
* Subjects who are judged ineligible for the clinical study by the investigator due to reasons other than the above inclusion/exclusion criteria.

Ages: 19 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Up to Post Study Visit (Part I SAD: Day 7~Day 9/ Part I SAD, FES: Day 14~ Day 16/ Part II:Day 13~Day 15)
  For all adverse events collected during the study, the investigator will evaluate serious adverse events, severity, or drug relationship
Vital Sign | Part I : Up to Day 3/ Part II: Up to Day 9
  Vital sign results will be classified as normal, not clinically significant, or clinically significant upon judgment of the investigator after single/multiple dosing of IN-114199
Physical Examination | Part I : Up to Day 3/ Part II: Up to Day 9
  Physical examination results will be classified as normal, not clinically significant, or clinically significant upon a judgment of the investigator after single/multiple dosing of IN-114199.
Body Weight in kilograms Measurement | Part I : Up to Day 3 / Part II: Up to Day 9
  The body weight in kilograms of Subjects will be monitored daily from the administration of IN-114199 until their discharge
12-lead electrocardiogram (ECG) | Part I SAD: Up to Day 3 / Part II: Up to Day 9
  QT/QTc interval will be recorded and analyzed automatically.
Clinical Laboratory Test | Part I:Day 1, Day 3/ Part II: Day 1, Day 3, Day 5, Day 7, Day 9
  Clinical laboratory test, the results will be classified as normal, not clinically significant, or clinically significant upon judgment of the investigator after single/multiple dosing of IN-114199

SECONDARY OUTCOMES:
PK parameters (Urine and Plasma) | Part I SAD: Up to Day 3/ Part I SAD, FES: Up to Day 3 / Part II: Up to Day 9
  Cmax
PK parameters (Urine and Plasma) | Part I SAD: Up to Day 3/ Part I SAD, FES: Up to Day 3 / Part II: Up to Day 9
  AUClast
PD parameters (plasma C4 level) | Part I SAD: Up to Day 3/ Part I SAD, FES: Up to Day 3 / Part II: Up to Day 9
  AUEClast
PD parameters (plasma LDL/HDL level) | Part I SAD: Up to Day 2/ Part I SAD, FES: Up to Day 2 / Part II: Up to Day 8
  AUEClast

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea